CLINICAL TRIAL: NCT00146575
Title: Randomized Trial of Paclitaxel-Eluting Stent and Sirolimus-Eluting Stent for Restenosis Reduction in Small Coronary Vessels (ISAR-SMART-3)
Brief Title: Sirolimus- and Paclitaxel-Eluting Stents for Small Vessels (ISAR-SMART-3)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S01703
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): randomized patients get sirolimus stent
  Interventions: Device: Sirolimus-eluting stent (Cypher)
- 2 (Experimental): randomized patients get paclitaxel stent
  Interventions: Device: Paclitaxel-eluting stent (Taxus)

INTERVENTIONS:
Device: Sirolimus-eluting stent (Cypher) — patients have been implanted a Cypher stent
  Other Names: Cypher
  Arms: 1
Device: Paclitaxel-eluting stent (Taxus) — patients have been implanted a Taxus stent
  Other Names: Taxus
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy of paclitaxel- and sirolimus-eluting stents to prevent re-blockage of small coronary arteries

DETAILED DESCRIPTION:
Although use of bare metal stents has reduced restenosis in coronary vessels with a diameter ≥3 mm when compared to plain balloon angioplasty, most of the dedicated randomized studies have failed to show a beneficial effect of stent over balloon angioplasty in vessels with a small reference diameter. In spite of refinements in stent design and periprocedural therapy, the risk of restenosis after bare metal stenting in this setting remains elevated. Nowadays, percutaneous coronary interventions in small vessels account for 35-67% of interventional procedures performed in patients with coronary artery disease and, when bare metal stents are used, restenosis will be detected in more than 35% of the treated patients and a repeat revascularization procedure will be needed in more than 20% them. Several randomized trials have shown that stents eluting antiproliferative drugs, with sirolimus- and paclitaxel-eluting stents the only devices approved for commercial use so far, are highly effective in reducing restenosis when compared with bare metal stents. Subgroup analysis from these trials have shown that the efficacy of either sirolimus stent or paclitaxel stent extends also to those patients who undergo coronary stenting in small sized vessels. In addition, three randomized studies of sirolimus-eluting stents and bare metal stents used in coronary arteries smaller than 3 mm have reported 82-96% reduction in the relative risk of restenosis with the sirolimus stents thus, providing convincing evidence on the role of drug-eluting stents as an effective treatment strategy for coronary arteries with a small reference diameter.

At present, there is no direct evidence on the relative efficacy in the prevention of restenosis of sirolimus stent and paclitaxel stent after implantation in small coronary vessels. Selecting the most effective device for this particularly high-risk category that accounts for a large proportion of percutaneous coronary interventions, may have important clinical and economic implications. Comparisons of data from subgroup analysis of different trials have suggested that there might be differences in the efficacy to prevent restenosis between sirolimus and paclitaxel stents. However, indirect comparisons are subject to many limitations and consequently, conclusions based on their results may be erroneous. Therefore, reliable guidance on the selection of the most effective drug-eluting stent for treatment of lesions in coronary vessels with a small reference diameter could be provided only from a head-to-head comparison between these devices.

Comparison:

Sirolimus-eluting stent and paclitaxel-eluting stent in patients undergoing stenting in small coronary vessels.

ELIGIBILITY:
Inclusion Criteria:

* Stable or unstable angina pectoris and/or a positive stress test
* "de novo" lesion in small coronary arteries (vessel size <2.8 mm by visual estimation)
* Written informed consent

Exclusion Criteria:

* Diabetes mellitus
* Myocardial infarction within 48 h. before enrollment
* Target lesion located in the left main trunk or bypass graft
* Contraindication or known allergy to aspirin, thienopyridines, rapamycin, paclitaxel or stainless steel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2003-06; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Late luminal loss | 6 months

SECONDARY OUTCOMES:
Binary angiographic restenosis | 1 year
Target lesion revascularization | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schomig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - Deutsches Herzzentrum, Munich

REFERENCES:
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Stone GW, Ellis SG, Cox DA, Hermiller J, O'Shaughnessy C, Mann JT, Turco M, Caputo R, Bergin P, Greenberg J, Popma JJ, Russell ME; TAXUS-IV Investigators. A polymer-based, paclitaxel-eluting stent in patients with coronary artery disease. N Engl J Med. 2004 Jan 15;350(3):221-31. doi: 10.1056/NEJMoa032441. PMID 14724301
- [Background] Kastrati A, Dibra A, Eberle S, Mehilli J, Suarez de Lezo J, Goy JJ, Ulm K, Schomig A. Sirolimus-eluting stents vs paclitaxel-eluting stents in patients with coronary artery disease: meta-analysis of randomized trials. JAMA. 2005 Aug 17;294(7):819-25. doi: 10.1001/jama.294.7.819. PMID 16106007
- [Background] Morice MC. Stenting for small coronary vessels. J Invasive Cardiol. 2003 Jul;15(7):377-9. No abstract available. PMID 12840233
- [Result] Mehilli J, Dibra A, Kastrati A, Pache J, Dirschinger J, Schomig A; Intracoronary Drug-Eluting Stenting to Abrogate Restenosis in Small Arteries (ISAR-SMART 3) Study Investigators. Randomized trial of paclitaxel- and sirolimus-eluting stents in small coronary vessels. Eur Heart J. 2006 Feb;27(3):260-6. doi: 10.1093/eurheartj/ehi721. Epub 2006 Jan 9. PMID 16401670